CLINICAL TRIAL: NCT00500656
Title: Randomised Double Blind, Controlled, Parallel Group, Multicentre Study of a Subcutaneous Formulation of Icatibant Versus Oral Tranexamic Acid for the Treatment of Hereditary Angioedema (HAE)
Brief Title: Subcutaneous Treatment With Icatibant for Acute Attacks of Hereditary Angioedema (HAE)
Acronym: FAST2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JE049 #2102; 2004-001540-71 (EudraCT Number)
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Randomized controlled -Icatibant (Experimental): Subjects received S.C icatibant+ oral placebo
  Icatibant Form: solution for injection, 3 mL, 10 mg/mL Single dose: 30 mg (3 mL)
  Placebo Form: hard capsule Single dose: 2 capsules Frequency: 3 x 2 capsules for 2 days, taken orally, 6 to 8 hours apart
  Interventions: Drug: Icatibant; Drug: Oral Placebo
- Randomized controlled-Tranexamic acid (Active Comparator): Subjects received oral Tranexamic acid+ S.C. placebo
  Tranexamic acid Form: over encapsulated film tablet Single dose: 1000 mg (2 capsules) Frequency: 3 x 2 capsules for 2 days, taken orally, 6 to 8 hours apart
  Placebo Form: solution for injection, matched to icatibant for injection Single dose: 3 mL Frequency: one subcutaneous injection in the abdominal region
  Interventions: Drug: Tranexamic Acid; Drug: S.C. Placebo
- Controlled Open-label / laryngeal attack (Experimental): Patients with laryngeal symptoms at the baseline were not randomised but treated with icatibant open label during the controlled phase.
  Interventions: Drug: Icatibant
- Untreated patients at the baseline (Experimental): Patients who were screened and found eligible but did not experience an angioedema attack, or had an attack that was not severe enough to merit treatment while the controlled phase was ongoing were treated in the open label phase with icatibant
  Interventions: Drug: Icatibant

INTERVENTIONS:
Drug: Icatibant — Icatibant: a stable, synthetic decapeptide and specific BK B2 receptor antagonist.
  Other Names: Brand name, Firazyr®
  Arms: Controlled Open-label / laryngeal attack; Randomized controlled -Icatibant; Untreated patients at the baseline
Drug: Tranexamic Acid — over encapsulated film tablet an anti-fibrinolytic agent,is used in some European countries for the treatment of acute oedema episodes and the continuous prophylaxis of HAE.
  Arms: Randomized controlled-Tranexamic acid
Drug: Oral Placebo — hard capsule matched to tranexamic acid
  Other Names: Placebo
  Arms: Randomized controlled -Icatibant
Drug: S.C. Placebo — solution for injection, matched to icatibant for injection
  Other Names: Placebo
  Arms: Randomized controlled-Tranexamic acid

SUMMARY:
Primary Outcome Measures:

The primary endpoint was the time to onset of symptom relief of the first attack in the double blind phase. H0: λ icatibant/λ tranexamic acid =1 versus H1: λ icatibant/λ tranexamic acid ≠1 Where: λ icatibant refers to the hazard rate under icatibant and λ tranexamic acid refers to the hazard rate under tranexamic acid.

Secondary Outcome Measures:

* Additional efficacy assessments (Time to Almost Complete Symptom Relief)
* Safety and tolerability
* Pharmacoeconomics

DETAILED DESCRIPTION:
This was a Phase III, randomised, double blind, double dummy, multicentre, controlled,parallel group study of a 30 mg s.c. formulation of icatibant for the treatment of patients with moderate to very severe symptoms of cutaneous and/or abdominal symptoms of HAE.

The study consisted of two parts: controlled phase and OLE phase. For the primary endpoint, Efficacy was determined by evaluating the differences in study outcomes using a Visual Analogue Scale for patients treated with icatibant and tranexamic acid.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years;
* Documented diagnosis of HAE Type I or II (confirmed C1-INH deficiency);
* Current edema in the cutaneous, abdominal and/or laryngeal areas;
* Current edema moderate to severe according to the investigator's Symptom Score.

Exclusion Criteria:

* Diagnosis of angioedema other than HAE,
* Participation in a clinical trial of another investigational medicinal product (IMP)within the past month
* Treatment with any pain medication since onset of the current angioedema attack
* Treatment with replacement therapy, including C1-INH products, less than 3 days before onset of the current angioedema attack
* Treatment with Tranexamic acid replacement therapy within a week before onset of the current angioedema attack
* Treatment with ACE inhibitors
* Contraindications for Tranexamic acid
* Evidence of coronary artery disease based on medical history or Screening examination in particular unstable angina pectoris or severe coronary heart disease
* Congestive heart failure (class 3 and 4)
* Serum creatinine level of ≥ 250 μmol/L
* Serious concomitant illness that the investigator considered to be a contraindication for participation in the trial
* Pregnancy (as assessed prior to treatment) and/or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2006-07-25 (Actual); Study Completion 2006-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Università degli Studi di Milano, Dipartimento di Medicina Interna, Milan, Italy

REFERENCES:
- [Result] Bas M, Bier H, Greve J, Kojda G, Hoffmann TK. Novel pharmacotherapy of acute hereditary angioedema with bradykinin B2-receptor antagonist icatibant. Allergy. 2006 Dec;61(12):1490-2. doi: 10.1111/j.1398-9995.2006.01197.x. No abstract available. PMID 17073887
- [Derived] Bas M, Greve J, Hoffmann TK, Reshef A, Aberer W, Maurer M, Kivity S, Farkas H, Floccard B, Arcoleo F, Martin L, Sitkauskiene B, Bouillet L, Schmid-Grendelmeier P, Li H, Zanichelli A. Repeat treatment with icatibant for multiple hereditary angioedema attacks: FAST-2 open-label study. Allergy. 2013 Nov;68(11):1452-9. doi: 10.1111/all.12244. Epub 2013 Sep 21. PMID 24111645
- [Derived] Cicardi M, Banerji A, Bracho F, Malbran A, Rosenkranz B, Riedl M, Bork K, Lumry W, Aberer W, Bier H, Bas M, Greve J, Hoffmann TK, Farkas H, Reshef A, Ritchie B, Yang W, Grabbe J, Kivity S, Kreuz W, Levy RJ, Luger T, Obtulowicz K, Schmid-Grendelmeier P, Bull C, Sitkauskiene B, Smith WB, Toubi E, Werner S, Anne S, Bjorkander J, Bouillet L, Cillari E, Hurewitz D, Jacobson KW, Katelaris CH, Maurer M, Merk H, Bernstein JA, Feighery C, Floccard B, Gleich G, Hebert J, Kaatz M, Keith P, Kirkpatrick CH, Langton D, Martin L, Pichler C, Resnick D, Wombolt D, Fernandez Romero DS, Zanichelli A, Arcoleo F, Knolle J, Kravec I, Dong L, Zimmermann J, Rosen K, Fan WT. Icatibant, a new bradykinin-receptor antagonist, in hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):532-41. doi: 10.1056/NEJMoa0906393. PMID 20818888

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 85 patients participated in the study(36 in the icatibant group and 38 in the tranexamic acid group)3 patients with laryngeal symptoms at Baseline.8 Patients were screened and found eligible but did not experience an angioedema attack, or had an attack that was not severe enough to merit treatment while the controlled phase was ongoing
Groups:
- Randomized Controlled -Icatibant: Patients who were randomized to icatibant + Oral placebo (hard capsule matched to tranexamic acid) in the controlled phase after they had an eligible first in-study attack.
- Randomized Controlled-Tranexamic Acid: Patients who were randomized to received oral Tranexamic acid + S.C. placebo(solution for injection, matched to icatibant for injection) in the controlled phase after they had an eligible first in-study attack.
Period: Controlled Phase
Arm/Group | Randomized Controlled -Icatibant | Randomized Controlled-Tranexamic Acid | Controlled Open-label / Laryngeal Attack | Untreated Patients at the Baseline
Started | 36 | 38 | 3 | 8
Completed | 26 | 28 | 2 | 0
Not Completed | 10 | 10 | 1 | 8
Period: Open Label Extension (OLE) Phase
Arm/Group | Randomized Controlled -Icatibant | Randomized Controlled-Tranexamic Acid | Controlled Open-label / Laryngeal Attack | Untreated Patients at the Baseline
Started | 23 (3 Subjects did not experience an angioedema attack after their first attack in the controlled phase) | 21 (7 Subjects did not experience an angioedema attack after their first attack in the controlled phase) | 2 | 8 (Subjects did not experience an angioedema attack during the controlled phase)
Completed | 16 | 9 | 1 | 6
Not Completed | 7 | 12 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Controlled -Icatibant | Randomized Controlled-Tranexamic Acid | Controlled Open-label / Laryngeal Attack | Untreated Patients at the Baseline | Total
Number analyzed (Participants) | 36 | 38 | 3 | 8 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (13.59) | 41.9 (12.36) | 35.0 (11.36) | 40.6 (13.51) | 40.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 1 | 7 | 55
  Male | 12 | 15 | 2 | 1 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 3 | 4 | 0 | 1 | 8
  France | 3 | 1 | 0 | 2 | 6
  Germany | 13 | 12 | 0 | 0 | 25
  Hungary | 3 | 3 | 0 | 0 | 6
  Ireland | 0 | 1 | 0 | 0 | 1
  Israel | 4 | 4 | 3 | 4 | 15
  Italy | 3 | 5 | 0 | 1 | 9
  Lithuania | 1 | 2 | 0 | 0 | 3
  Poland | 1 | 2 | 0 | 0 | 3
  Sweden | 3 | 2 | 0 | 0 | 5
  Switzerland | 2 | 2 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Symptom Relief.
Description: The primary efficacy endpoint was Time to onset of symptom relief (TOSR) following treatment with either icatibant or tranexamic acid. The median time to onset of symptom relief for the icatibant group was compared to the the median time to onset of symptom relief for the tranexamic acid group. TOSR was defined as the time between time of injection to time of first documented onset of symptom relief for the three primary symptoms: cutaneous swelling, cutaneous skin, and abdominal pain. The primary symptom was based on the type of attack. For abdominal attacks, the single primary symptom was abdominal pain. For cutaneous attacks, the single primary symptom was either skin swelling or skin pain, whichever was most severe.
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Randomized Controlled -Icatibant | Randomized Controlled-Tranexamic Acid
Number analyzed (Participants) | 36 | 38
Hours | 2.0 [1.0 to 3.5] | 12.0 [3.5 to 25.4]
Statistical Analysis 1: Comparison: Randomized Controlled -Icatibant vs Randomized Controlled-Tranexamic Acid; Test type: Superiority or Other; p < 0.001, The Wilcoxon version of the log rank; The median time to onset was calculated using Kaplan Meier methodology. The Wilcoxon version of the log rank test of SAS was used; Hazard Ratio (HR) = 3.475, 95% CI 2-sided [1.901 to 6.355]

2. Secondary Outcome: Time to Almost Complete Symptom Relief
Description: Almost complete symptom relief was defined as a score between 0 and 10 mm on the VAS for at least three consecutive measurements for all symptoms.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Randomized Controlled -Icatibant | Randomized Controlled-Tranexamic Acid
Number analyzed (Participants) | 36 | 38
Hours | 10.0 [2.8 to 23.2] | 51.0 [12.0 to 79.5]
Statistical Analysis 1: Comparison: Randomized Controlled -Icatibant vs Randomized Controlled-Tranexamic Acid; Test type: Superiority or Other; p < 0.001, The Wilcoxon version of the log rank; The median time to almost complete symptom relief was calculated using Kaplan Meier methodology.The Wilcoxon version of the log rank test SAS was used

ADVERSE EVENTS:
Time Frame: An AE was assigned to the controlled phase if the start date of the event was between the first treatment of the first attack and the first treatment in the OLE phase.
Groups:
- Controlled Phase- Icatibant (Randomized Subjects ): Patients who were randomized to icatibant+ oral placebo in the controlled phase and experienced adverse events while participating in the controlled phase
- Controlled Phase- Tranexamic Acid (Randomized Subjects): Patients who were randomized to Tranexamic acid+ S.C. placebo in the controlled phase and experienced adverse events while participating in the controlled phase.
- Controlled Phase- Icatibant (Subjects w/ Laryngeal Attack): This represents adverse events during the controlled phase that were experienced by Patients with laryngeal symptoms at the baseline and were treated with open label icatibant during the controlled phase.
- Open Label Extension Phase- Icatibant (Previously Randomized): Patients who were randomized to either icatibant+ oral placebo or Tranexamic acid+ S.C. placebo in the controlled phase and experienced adverse events while participating in the open label extension phase.
- Open Label Extension Phase (Subjects w/ Laryngeal Attack): This represents adverse events during the open label extension phase that were experienced by Patients with laryngeal symptoms at the baseline and got treated with open label icatibant during the controlled phase and Open label extension phase.
- Open Label Extension Phase(Untreated Patients at the Baseline: This represents adverse events experienced by Patients who were screened and found eligible but did not experience an angioedema attack, or had an attack that was not severe enough to merit treatment while the controlled phase was ongoing.
Arm/Group | Controlled Phase- Icatibant (Randomized Subjects ) | Controlled Phase- Tranexamic Acid (Randomized Subjects) | Controlled Phase- Icatibant (Subjects w/ Laryngeal Attack) | Open Label Extension Phase- Icatibant (Previously Randomized) | Open Label Extension Phase (Subjects w/ Laryngeal Attack) | Open Label Extension Phase(Untreated Patients at the Baseline
Serious Adverse Events (participants affected / at risk) | 4/36 | 1/38 | 1/3 | 9/44 | 1/2 | 0/8
Other Adverse Events (participants affected / at risk) | 19/36 | 16/38 | 1/3 | 31/44 | 1/2 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Controlled Phase- Icatibant (Randomized Subjects ) (N=36) | Controlled Phase- Tranexamic Acid (Randomized Subjects) (N=38) | Controlled Phase- Icatibant (Subjects w/ Laryngeal Attack) (N=3) | Open Label Extension Phase- Icatibant (Previously Randomized) (N=44) | Open Label Extension Phase (Subjects w/ Laryngeal Attack) (N=2) | Open Label Extension Phase(Untreated Patients at the Baseline (N=8)
Hereditary Angioedema (Congenital, familial and genetic disorders) | 2 | 0 | 1 | 3 | 1 | 0
Aortic Value Sclerosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sudden Cardiac Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic Enzymes Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Urinary Track Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Controlled Phase- Icatibant (Randomized Subjects ) (N=36) | Controlled Phase- Tranexamic Acid (Randomized Subjects) (N=38) | Controlled Phase- Icatibant (Subjects w/ Laryngeal Attack) (N=3) | Open Label Extension Phase- Icatibant (Previously Randomized) (N=44) | Open Label Extension Phase (Subjects w/ Laryngeal Attack) (N=2) | Open Label Extension Phase(Untreated Patients at the Baseline (N=8)
Hereditary Angioedema (Congenital, familial and genetic disorders) | 10 | 6 | 1 | 10 | 1 | 1
Injection Site Reaction (General disorders) | 2 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3 | 0 | 4 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0
Urinary Track Infection (Infections and infestations) | 0 | 0 | 0 | 6 | 0 | 0
Gingival Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dental Caries (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Track Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dental Operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Blood and Lymphatic system disorders (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 0 | 0
Injury, poisoning and procedual complications (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 3 | 0 | 0
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less